CLINICAL TRIAL: NCT04116996
Title: Stimulation of the External Pallidal Segment for Insomnia in Patients With Parkinson's Disease
Brief Title: Globus Pallidus Stimulation to Treat Insomnia
Acronym: GPS-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Pablo Castillo, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-010112
Record Dates: First submitted 2019-10-02; First posted 2019-10-07 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Adults with Parkinson's disease and severe insomnia (Experimental): 1 arm study
  Interventions: Device: DEEP BRAIN STIMULATION

INTERVENTIONS:
Device: DEEP BRAIN STIMULATION — NEUROMODULATION

SUMMARY:
Researchers are to determine if turning on an additional unilateral DBS (deep brain stimulation) electrode with stimulation to the globus pallidus externa (GPe) region of the brain will improve insomnia (sleep).

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years of age
* Symptomatic with Parkinsonism for 7-20 years
* Severe insomnia based on ISI score

Exclusion Criteria:

* Clinically significant dementia (MMSE <23)
* Hoehn & Yahr [Hoehn, 1967 #1839] stage I or V disease
* Other significant neurological or psychiatric disease
* Previous pallidotomy or thalamotomy
* Previous placement of other implantable devices
* Secondary parkinsonism (non-idiopathic parkinsonism)
* Inability to travel to Jacksonville for post-operative study visits
* Severe sleep apnea
* Insomnia due to pain or untreated mood disorder
* Contraindications to 3T MRI
* Circadian rhythm sleep disorders.
* Current use of hypnotics

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | 3 and 6 months
  Change in self-reported insomnia severity index questionnaire score, using a total score scale of 0-7 is no clinically significant insomnia, 8-14 is subthreshold insomnia, 15-21 is clinical insomnia (moderate severity), 22-28 is Clinical insomnia (severe)

SECONDARY OUTCOMES:
Change in Parkinson's Sleep Scale (PDSS) | 3 and 6 months
  Change in self-reported Parkinson's Sleep Scale (PDSS) questionnaire, using a scale of 0 is always and 10 as never

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Castillo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials